CLINICAL TRIAL: NCT04728009
Title: Safety and Efficacy of Longan and Lingzhi Mushroom Syrup on Immune and Inflammatory Responses in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REH-62320
Record Dates: First submitted 2020-12-23; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- longan and lingzhi mushroom syrup (Experimental): All participants (N = 8) were asked to consume 5 mL of longan and lingzhi mushroom syrup as a sweetener daily for 12 weeks.
  Interventions: Dietary Supplement: Longan and lingzhi mushroom syrup

INTERVENTIONS:
Dietary Supplement: Longan and lingzhi mushroom syrup — Fresh fruit pulps of longan were stewed in hot water until they softened. No sugar and additives were added. The pulps were removed by filtration in order to obtain concentrated longan juice. After that, spray-dried powder of lingzhi mushroom extract was dissolved in water in the ratio of 1:2. To make the finished product, 99 g of longan juice was mixed with 1 g of the lingzhi extract in water. The sugar content of the syrup was 77 degrees Brix.

SUMMARY:
This study aimed to preliminarily determine safety and efficacy of longan and lingzhi mushroom syrup on immune and inflammatory responses. Apparently healthy Thai adults (N = 8) aged 18-60 years were recruited into a prospective, single-group study. All participants were assigned to consume 5 mL of longan and lingzhi mushroom syrup daily for 12 weeks. Blood concentrations of fasting plasma glucose (FPG), glycated hemoglobin (HbA1c), aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), BUN (blood urea nitrogen), creatinine (Cr), immunoglobulins (IgG, IgM, IgA, and IgE), and C-reactive protein (CRP) were measured at baseline (week 0), week 4, week 8, and week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy adults at Mae Fah Luang University and Chulalongkorn University
2. aged 18-60 years
3. HbA1c < 7%

Exclusion Criteria:

1. self-reported immunodeficiency diseases, autoimmune diseases, infectious diseases, diabetes, thyroid diseases, cancer, hepatic- and/or renal dysfunction, uncontrollable illnesses and life-threatening diseases
2. being allergic to longan and lingzhi products
3. taking medications, herbs, and diet supplements affecting immune system, inflammatory response, and blood glucose a month before study enrollment
4. pregnant and breastfeeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Adverse effects on fasting blood glucose | 12 weeks
  Blood concentrations of fasting blood glucose (in mg/dL) were measured.
Adverse effects on long-term glycemic control | 12 weeks
  Blood concentrations of HbA1C (in %) were measured.
Adverse effects on hepatic function (1) | 12 weeks
  Blood concentrations of aspatate aminotransferase (AST) (in units/L) were measured.
Adverse effects on hepatic function (2) | 12 weeks
  Blood concentrations of alanine aminotransferase (ALT) (in units/L) were measured.
Adverse effects on hepatic function (3) | 12 weeks
  Blood concentrations of alkaline phosphatase (ALP) (in units/L) were measured.
Adverse effects on renal function (1) | 12 weeks
  Blood concentrations of blood urea nitrogen (in mg/dL) were measured.
Adverse effects on renal function (2) | 12 weeks
  Blood concentrations of serum creatinine (in mg/dL) were measured.

SECONDARY OUTCOMES:
Effect on immune responses (1) | 12 weeks
  Blood concentrations of immunoglobulin (Ig) G (in mg/dL) were measured.
Effect on immune responses (2) | 12 weeks
  Blood concentrations of Ig M (in mg/dL) were measured.
Effect on immune responses (3) | 12 weeks
  Blood concentrations of Ig A (in mg/dL) were measured.
Effect on immune responses (4) | 12 weeks
  Blood concentrations of Ig E (in IU/mL) were measured.
Effect on inflammatory responses | 12 weeks
  Blood concentrations of C-reactive protein (in mg/L) were measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Thailand